CLINICAL TRIAL: NCT02965326
Title: Personalized Therapy of Cystic Fibrosis: Set-up of Response Markers
Brief Title: Surrogate Markers of Response to New Therapies in Cystic Fibrosis Patients
Acronym: BIO-CFTR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Necker-Enfants Malades (Other)
Collaborators: Association Mucoviscidose-ABCF2 (Other); Vaincre la Mucoviscidose (Other)
Responsible Party: Principal Investigator, Isabelle Sermet-Gaudelus, Professor, Hôpital Necker-Enfants Malades
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ABCF-2016-01; 2016-A00309-42 (Other: ANSM, French national agency for drug safety)
Record Dates: First submitted 2016-11-11; First posted 2016-11-16 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cystic fibrosis, treated (Other): Cystic fibrosis patients treated either by Ivacaftor or by the association Ivacaftor-Lumacaftor
  Interventions: Procedure: Nasal swab; rectal biopsy.
- Cystic fibrosis, non treated (Other): Cystic fibrosis patients, non treated by a CFTR modulator
  Interventions: Procedure: Nasal swab; rectal biopsy.
- Non-Cystic fibrosis (Other): Patients in whom cystic fibrosis diagnosis has been suspected, but excluded by physiological and genetic investigations
  Interventions: Procedure: Nasal swab; rectal biopsy.

INTERVENTIONS:
Procedure: Nasal swab; rectal biopsy. — Nasal epithelial cells will be obtained by nasal swabs from patients of the three arms; intestinal epithelial cells will be obtained, by rectal biopsy, only from patients treated by CFTR modulators.

SUMMARY:
The purpose of this study is to determine which biological marker, or association of biological markers, best predict clinical response of cystic fibrosis patients to CFTR modulators.

DETAILED DESCRIPTION:
This study is based upon the hypothesis that clinical response of cystic fibrosis patients to CFTR modulators is correlated to in vitro responses to these drugs of epithelial cells derived from the patients, as assessed by CFTR-dependent Chloride secretion. Epithelial cells will be derived either from nasal or rectal epithelia, and consist both of cultured cells and organoids. The drugs tested will be Ivacaftor, or Lumacaftor/Ivacaftor, according to patient's treatment. Results of these assays will be compared with response to treatment at 6 and 12 months, assessed by clinical response and in vivo assay of CFTR function.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis patients treated by CFTR modulators (Ivacaftor or the association Ivacaftor-Lumacaftor)
* Cystic fibrosis patients non treated by CFTR modulators
* Patients in whom cystic fibrosis diagnosis has been suspected, but excluded by physiological and genetic investigations

Exclusion Criteria:

* pregnant or lactating women
* contraindication to nasal swab
* contraindication to rectal biopsy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second | initiation, 7 days, 1 month, 6 months, 1 year and every 6 months
  Respiratory Function test

SECONDARY OUTCOMES:
Forced Vital Capacity | initiation, 7 days, 1 month, 6 months, 1 year and every 6 months
  Respiratory Function test
Forced Expiratory Flow 25-75 | initiation, 7 days, 1 month, 6 months, 1 year and every 6 months
  Respiratory Function test
Residual Volume | initiation, 7 days, 1 month, 6 months, 1 year and every 6 months
  Respiratory Function test
elastase in sputum | initiation, 7 days, 1 month, 6 months, 1 year and every 6 months
  elastase activity in UI/g of sputum
calprotectin in sputum | initiation, 7 days, 1 month, 6 months, 1 year and every 6 months
  calprotectin in µg/g of sputum
IL-8 in sputum | initiation, 7 days, 1 month, 6 months, 1 year and every 6 months
  IL-8 in µg/g of sputum
Calprotectin in blood | initiation, 1 month, 3 Months, 6 months and every 6 months
  calprotectin in µg/ml of blood
IL-8 in blood | initiation, 1 month, 3 Months, 6 months and every 6 months
  IL-8 in µg/ml of blood
tumor necrosis factor in sputum | initiation, 1 month, 3 Months, 6 months and every 6 months
  tumor necrosis factor in µg/g of sputum
liver function test in blood | initiation, 1 month, 3 Months, 6 months and every 6 months
  serum glutamate oxaloacetate transaminase in ui/ml
liver function test/SGPT in blood | initiation, 1 month, 3 Months, 6 months and every 6 months
  serum glutamate pyruvate transaminase in ui/ml
liver function test/bilirubin in blood | initiation, 1 month, 3 Months, 6 months and every 6 months
  Bilirubin in mg/ml
liver function test, gammaGT in blood | initiation, 1 month, 3 Months, 6 months and every 6 months
  GammaGT in UI/ml
creatine phosphokinase in blood | initiation, 1 month, 3 Months, 6 months and every 6 months
  CPK in mg/ml
Amylase in blood | initiation, 1 month, 3 Months, 6 months and every 6 months
  amylase in mg/ml
Impedancemetry | initiation , 1 month, 3 Months, 6 months and every 6 months
  ambulatory measurement of body composition
Dynamometry | initiation , 1 month, 3 Months, 6 months and every 6 months
  ambulatory measurement of quadriceps strength
Sweat test | initiation ,1 month
  chloride concentration in sweat
proteomics of sweat | initiation, 7 days, 1 month, 6 months, 1 year and every 6 months
  measurement of proteins in sweat
metabolomics of sweat | initiation, 7 days, 1 month, 6 months, 1 year and every 6 months
  measurement of métabolites in sweat
proteomics of exhalate | initiation, 7 days, 1 month, 6 months, 1 year and every 6 months
  measurement of proteins in exhaled air
sputum bronchial microorganism colonization | initiation , 1 month, 3 Months, 6 months and every 6 months
  bacterial, fungi and viral colonization
Lung MRI | initiation, at 1 year and every year
  Lung Imaging evaluation : number of bronchiectasis, number of mucus plugs
osteodensitometry | initiation, 1 year, and every year
  Bone mineralization body composition
fecal elastase | initiation, at 6 months and every year
  elastase feces in µg/g feces
fecal calprotectin | initiation, at 6 months and every year
  calprotectin, concentraion in feces in µg/g
Chest CT scan | initiation, 3 years and 5 years
  Lung Imaging: % versuys normal of lung parenchuma with bronchiectasis, airway wall thickening, mucus plugs, air trapping
glycemic Holter | initiation, 1 year and every year
  glycemia monitoring
abdominal ultrasonography | treatment initiation, 1 year and every year
  presence of liver hyperechogenicity, fibrosis, as assessed by the radiologist
proton density fat fraction | treatment initiation, 1 year
  magnetic resonance Imaging of the Pancreas
patient quality of life | initiation, 1 month, 6 months, 1 year and every 6 months
  Score tolerance of the treatment, perception of respiratory, digestive symptoms, energy, body image as assessed by the "Cystic Fibrosis Questionnaire" score a better quality of life is indicated by an increase in the score value. Minimum value is 0, maximum is 100.
CFTR activity in nasal cells/chloride | initiation of treatment and repeated if cell culture failure
  Chloride transport in primary nasal cell cultures obtained by nasal brushing and study in Ussing chamber (µA/cm2)
CFTR activity in nasal cells/bicarbonat | initiation of treatment and repeated if cell culture failure
  Bicarbonate transport in primary nasal cell cultures obtained by nasal brushing and study in Ussing chamber (µA/cm2)
CFTR activity in intestinal epithelium/chloride | initiation of treatment and repeated of cell culture failure
  Chloride transport in intestinal primary culture and study in Ussing chamber (µA/cm2)
CFTR activity in intestinal epithelium/bicarbonate | initiation of treatment and repeated of cell culture failure
  Bicarbonate transport in intestinal primary culture and study in Ussing chamber (µA/cm2)
sweat evaporimetry | initiation and 1 month
  quantity of sweat produced afer bet-adrenergic stimulation after subcutaneous injection
Elasto MRI | initiation and 1 year
  measurement of liver fibrosis by MRI
Lung Clearance Index | initiation, 6 months, 1 year and every 6 months
  Capacity of the lung to washout pure Oxygen,
proteomics in blood | initiation, 7 days, 1 month, 6 months, 1 year and every year
  measurement of proteins in blood
metabolomics in blood | initiation, 7 days, 1 month, 6 months, 1 year and every year
  measurement of métabolites in blood
proteomic in urine | initiation, 7 days, 1 month, 6 months, 1 year and every year
  measurement of proteins in blood
metabolomics in urine | initiation, 7 days, 1 month, 6 months, 1 year and every year
  measurement of métabolites in urine
Exhaled air composition | initiation, 7 days, 1 month, 6 months, 1 year and every year
  Volatile organic compounds in exhaled air

CONTACTS AND LOCATIONS:
Overall Officials: Aleksander Edelman, phD, Study Director — APHP
Locations (1):
- Necker Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramsey BW, Davies J, McElvaney NG, Tullis E, Bell SC, Drevinek P, Griese M, McKone EF, Wainwright CE, Konstan MW, Moss R, Ratjen F, Sermet-Gaudelus I, Rowe SM, Dong Q, Rodriguez S, Yen K, Ordonez C, Elborn JS; VX08-770-102 Study Group. A CFTR potentiator in patients with cystic fibrosis and the G551D mutation. N Engl J Med. 2011 Nov 3;365(18):1663-72. doi: 10.1056/NEJMoa1105185. PMID 22047557
- [Background] Graeber SY, Hug MJ, Sommerburg O, Hirtz S, Hentschel J, Heinzmann A, Dopfer C, Schulz A, Mainz JG, Tummler B, Mall MA. Intestinal Current Measurements Detect Activation of Mutant CFTR in Patients with Cystic Fibrosis with the G551D Mutation Treated with Ivacaftor. Am J Respir Crit Care Med. 2015 Nov 15;192(10):1252-5. doi: 10.1164/rccm.201507-1271LE. No abstract available. PMID 26568242
- [Background] Quittner A, Suthoff E, Rendas-Baum R, Bayliss MS, Sermet-Gaudelus I, Castiglione B, Vera-Llonch M. Effect of ivacaftor treatment in patients with cystic fibrosis and the G551D-CFTR mutation: patient-reported outcomes in the STRIVE randomized, controlled trial. Health Qual Life Outcomes. 2015 Jul 2;13:93. doi: 10.1186/s12955-015-0293-6. PMID 26135562
- [Background] De Boeck K, Munck A, Walker S, Faro A, Hiatt P, Gilmartin G, Higgins M. Efficacy and safety of ivacaftor in patients with cystic fibrosis and a non-G551D gating mutation. J Cyst Fibros. 2014 Dec;13(6):674-80. doi: 10.1016/j.jcf.2014.09.005. Epub 2014 Sep 26. PMID 25266159
- [Background] Boyle MP, Bell SC, Konstan MW, McColley SA, Rowe SM, Rietschel E, Huang X, Waltz D, Patel NR, Rodman D; VX09-809-102 study group. A CFTR corrector (lumacaftor) and a CFTR potentiator (ivacaftor) for treatment of patients with cystic fibrosis who have a phe508del CFTR mutation: a phase 2 randomised controlled trial. Lancet Respir Med. 2014 Jul;2(7):527-38. doi: 10.1016/S2213-2600(14)70132-8. Epub 2014 Jun 24. PMID 24973281
- [Background] Wainwright CE, Elborn JS, Ramsey BW, Marigowda G, Huang X, Cipolli M, Colombo C, Davies JC, De Boeck K, Flume PA, Konstan MW, McColley SA, McCoy K, McKone EF, Munck A, Ratjen F, Rowe SM, Waltz D, Boyle MP; TRAFFIC Study Group; TRANSPORT Study Group. Lumacaftor-Ivacaftor in Patients with Cystic Fibrosis Homozygous for Phe508del CFTR. N Engl J Med. 2015 Jul 16;373(3):220-31. doi: 10.1056/NEJMoa1409547. Epub 2015 May 17. PMID 25981758
- [Background] De Boeck K, Kent L, Davies J, Derichs N, Amaral M, Rowe SM, Middleton P, de Jonge H, Bronsveld I, Wilschanski M, Melotti P, Danner-Boucher I, Boerner S, Fajac I, Southern K, de Nooijer RA, Bot A, de Rijke Y, de Wachter E, Leal T, Vermeulen F, Hug MJ, Rault G, Nguyen-Khoa T, Barreto C, Proesmans M, Sermet-Gaudelus I; European Cystic Fibrosis Society Clinical Trial Network Standardisation Committee. CFTR biomarkers: time for promotion to surrogate end-point. Eur Respir J. 2013 Jan;41(1):203-16. doi: 10.1183/09031936.00057512. Epub 2012 Aug 9. PMID 22878883
- [Background] Dekkers JF, Wiegerinck CL, de Jonge HR, Bronsveld I, Janssens HM, de Winter-de Groot KM, Brandsma AM, de Jong NW, Bijvelds MJ, Scholte BJ, Nieuwenhuis EE, van den Brink S, Clevers H, van der Ent CK, Middendorp S, Beekman JM. A functional CFTR assay using primary cystic fibrosis intestinal organoids. Nat Med. 2013 Jul;19(7):939-45. doi: 10.1038/nm.3201. Epub 2013 Jun 2. PMID 23727931
- [Derived] Pranke I, Hatton A, Masson A, Flament T, Le Bourgeois M, Chedevergne F, Bailly C, Urbach V, Hinzpeter A, Edelman A, Sermet-Gaudelus I. Might Brushed Nasal Cells Be a Surrogate for CFTR Modulator Clinical Response? Am J Respir Crit Care Med. 2019 Jan 1;199(1):123-126. doi: 10.1164/rccm.201808-1436LE. No abstract available. PMID 30326728